CLINICAL TRIAL: NCT06356974
Title: An Intervention Study to Evaluate the Impact of Treating gHAT Seropositive Subjects With Acoziborole on Transmission of T.b. Gambiense, and Obtain Further Safety Data on Acoziborole in gHAT Seropositive Individuals
Brief Title: Stop Transmission of Gambiense Human African Trypanosomiasis (STROgHAT)
Acronym: STROgHAT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Institut de Recherche pour le Developpement (Other Government); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STROgHAT
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Human African Trypanosomiasis
Keywords: acoziborole, elimination of transmission, seropositive

STUDY DESIGN:
Intervention Model Description: one-arm, open label, non-randomized, multicentre, phase IIIb study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of seropositives (Experimental): * acoziborole three 320-mg tablets (960 mg dose), administered by the oral route to adolescent and adults ≥15 years as single dosing regimen on Day 1 of the study in fed or fasting state
  * acoziborole two 320-mg tablets (640 mg dose), administered by the oral route to children 11-14 years (and ≥30kg) as single dosing regimen on Day 1 of the study in fed or fasting state No active comparative treatment will be used in this study
  Doses and treatment regimens
  * Adolescent and adults ≥15 years: 960 mg (3x320mg) oral unique dose in fed or fasting state
  * Children 11-14 years (and ≥30kg): 640 mg (2x320mg) oral unique dose in fed or fasting state
  Interventions: Drug: Treatment of seropositive individuals (positive serology test, but parasitology not confirmed)

INTERVENTIONS:
Drug: Treatment of seropositive individuals (positive serology test, but parasitology not confirmed) — Subjects agreeing to participate in the study and matching the inclusion/exclusion criteria will receive acoziborole 960 or 640 mg in a single intake at study day 1. Following treatment, participants will attend follow-up visits at home or at the study centre at 3 days and 3-months post treatment.
  Other Names: Acoziborole

SUMMARY:
This protocol describes both the epidemiological study which aims at assessing whether over a three-year period a zero prevalence can be achieved when implementing a screen & treat approach with acoziborole, as well as a nested clinical study aimed at generating further evidence on safety of acoziborole in gambiense human African trypanosomiasis (gHAT) seropositives individuals. The overall coordinator will be ITM. ITM will be fully responsible for the epidemiological study (study Part A), including cost effectiveness and evaluation of diagnostic tests. DNDi will be the legal sponsor of the nested safety clinical study (study Part B) and will ensure compliance with regulatory requirements and good clinical practices (GCP) for this part of the study.

The investigators hypothesize that by systematically screening the populations of all endemic villages in a well-defined HAT focus and by expanding gHAT treatment to all seropositives, that it will be able to arrive at a zero prevalence over a three-year period.

The objectives are to evaluate whether a strategy based on widened treatment for all parasitologically negative seropositive gHAT suspects with acoziborole can lead to interruption of transmission of T.b.gambiense in a mainland focus and to assess the safety of acoziborole in gHAT seropositve individuals and parasitologically negative.

DETAILED DESCRIPTION:
Recently acoziborole, a non-toxic single dose oral drug for gHAT, has passed phase 3 evaluation in adult patients. This drug is envisioned to be used to treat gHAT irrespective of disease stage, thus rendering the lumbar puncture for stage determination redundant. Having available a single dose oral treatment with limited risk of toxicity opens up new perspectives for eliminating the disease. Treating anyone testing positive to a serological screening test, without further need for on the spot parasitological confirmation and stage determination, will greatly simplify procedures in the field, avoid missing many cases, has the potential to increase uptake of screening and may thus even curb transmission of the causative parasite, which is assumed to have only a human reservoir.

Although this innovative option for gHAT control is now feasible, its true effectiveness and cost effectiveness for curtailing transmission remain to be determined.

The current gHAT control strategy is based on active screening of people living in villages at risk for gHAT by mobile screening teams. All villages from which gHAT cases were reported are screened for three years in a row until no further cases are found. They are then screened once more, two years after the last case was reported. If no further cases are found, transmission is assumed to have been interrupted. However, it has also previously been shown estimated that up to 50% of prevalent cases are not detected or not cured, with major losses occurring during the parasitological confirmation step. Other important barriers are the fear of the lumbar puncture required for stage determination and of toxicity of treatment, in particular associated with melarsoprol, no longer in use for gHAT, but still well-known especially by the elder population. Even if up to 50% of prevalent gHAT cases were not treated, the epidemiological data shows that the disease is on the decline. This may however be insufficient to achieve complete elimination of transmission. The investigators hypothesize that by systematically screening the populations of all endemic villages in a well-defined HAT focus and by expanding gHAT treatment to all seropositives, that it will be able to arrive at a zero prevalence over a three-year period. Bearing in mind that acoziborole has not yet been registered and that 'screen & treat' has not yet been adopted as the new policy, the investigators will for the duration of this study continue performing parasitological confirmation on the spot and treat anyone confirmed by parasitology with standard of care. Any serological suspect not confirmed by parasitology on the spot will be offered treatment with acoziborole (study Part B), conditional on a set of inclusion and exclusion criteria If acoziborole allows the investigators to implement a screen & treat strategy, allowing to detect and treat all g-HAT prevalent cases, and possibly in the future without the limitations of cumbersome diagnostic confirmation on the spot, the investigators expect that elimination of transmission is also possible in a mainland focus. Implementing such a study under relatively well controlled conditions will also allow gathering further evidence on safety of acoziborole, before a screen & treat strategy is rolled out on a larger scale. In addition it will provide information on the cost of such a strategy and on some essential parameters of the tests utilized.

ELIGIBILITY:
Inclusion Criteria:

* • Participants able to give signed informed consent and assent form for adolescents, which includes willingness to comply with the schedule of follow-up visits and other requirements and restrictions listed in the informed consent form (ICF) and in this protocol

  * All sexes
  * 11 years of age or older at the start of the study and weight ≥30 kg at the screening of Part B
  * Participants who are CATT test or HAT RDT positive (information provided by the mobile team and included into TrypElim (see Part A)
  * Participants who are able to ingest oral tablets
  * Participants with known address and/or contact details provided
  * Participants who are able to comply with the schedule of follow-up visits and other requirements of the study
  * Participants must agree not take part in any other clinical trials during the participation in part B of this study
  * Participants of child-bearing potential must be willing to use appropriate contraceptive methods.

Exclusion Criteria:

* • Individuals with a positive parasitological exam on the spot at baseline (mAECT or lymph gland puncture)

  * Participants previously treated for g-HAT or previously treated because of gHAT seropositive results
  * Pregnant women
  * Breast-feeding women
  * Children ≥11 years, but under 30kg body weight at the screening for part B
  * Clinically significant medical condition that could, in the opinion of the investigator, jeopardise the subject's safety or participation in the study
  * Individuals presenting a jaundice at screening
  * Participants who are taking, or who are expected to need to start within 3 months, a medicine (including traditional or herbal) which may interact with acoziborole and which cannot be stopped or adjusted (please refer to investigator manual or contact DNDi)

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Interruption of transmission of T.b. gambiense | 4 years
  to evaluate whether a strategy based on widened treatment for all parasitologically negative seropositive gHAT suspects with Acoziborole can lead to interruption of transmission of HAT in a mainland focus The HAT prevalence with 95%CI will be calculated using the data from active and passive screening campaigns during year 1,2,3 of the project. Participation rate to the screening activities per age group and sex will also be calculated during the study period.
  The primary endpoint is the prevalence of confirmed HAT cases, either at point of care by parasitological tests or at the reference laboratory by a positive immunological test (ELISA/T.b.gambiense or trypanolyisi) AND a positive molecular test (18S rRNA or q177T). This prevalence will be determined among the population screened during the fourth and final survey round.
Assessment of safety | 3 years
  Proportion of participants who present related treatment emergent severe adverse events (severe related TEAEs) Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) SOC and PT. The primary endpoint for this study is the occurrence of severe related TEAEs from administration of study drug up to 3 months post-treatment. It is a binary endpoint (presence or absence of severe TEAE). Other safety endpoints will be collected and analyzed in the same manner as the primary endpoints.
  * Proportion of participants with mild or moderate related TEAES
  * Proportion of participants with any (mild, moderate, severe) TEAES
  * Proportion of participants with serious treatment emergent adverse events (TESAEs) from time of first administration

SECONDARY OUTCOMES:
Economic evaluation | 4 years
  Cost data will be gathered throughout the study and used to perform an economic evaluation of the screen & treat strategy in the study area. A separate analysis plan will be developed. The investigators will cost the strategy using a health-care provider's perspective, focusing on costs incurred by the Ministry of Health (PNLTHA and INRB) and donors. Only costs related to the STROGHAT elimination strategy will be considered, research and management costs will be excluded. A mixed costing methodology will be used to estimate financial and economic costs. Recurrent and capital costs will be considered. The sensitivity analysis will use discount rates of 0%, 5% and 10% and evaluate the impact of the main cost drivers. The cost information collected will also be used to develop a tool to support national programs estimate the cost and budget necessary if they would like to implement a similar intervention in a different context if the trial shows promising results.
assessment of the performance of several diagnostic tests | 4 years
  The specificity of the diagnostic tests used in the study: CATT and RDTs in the field, and ELISA/T.b. gambiense, immune trypanolysis and Trypanozoon-RT-PCR multiplex at INRB level, will be evaluated. The reference standard will be parasitological confirmation. The specificity of the different tests will be calculated by measuring the number of index tests négatives over the number of index test négatives plus index test positives tesing negative with the reference test.
  Senstivity will not be calculated as in the context of low prevalence, only few positives are detected not allowing for statistical inference.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Nicco, MD, Study Director — Institute of Tropical Medicine

IPD SHARING:
Plan to Share IPD: No
anonymity of participants must be guaranteed, GDRPR rules will apply anonymised study results can be shared with other researchers upon request

REFERENCES:
- [Background] Robays J, Bilengue MM, Van der Stuyft P, Boelaert M. The effectiveness of active population screening and treatment for sleeping sickness control in the Democratic Republic of Congo. Trop Med Int Health. 2004 May;9(5):542-50. doi: 10.1111/j.1365-3156.2004.01240.x. PMID 15117297
- [Background] Dickie EA, Giordani F, Gould MK, Maser P, Burri C, Mottram JC, Rao SPS, Barrett MP. New Drugs for Human African Trypanosomiasis: A Twenty First Century Success Story. Trop Med Infect Dis. 2020 Feb 19;5(1):29. doi: 10.3390/tropicalmed5010029. PMID 32092897
- [Background] Simarro PP, Cecchi G, Franco JR, Paone M, Diarra A, Ruiz-Postigo JA, Fevre EM, Mattioli RC, Jannin JG. Estimating and mapping the population at risk of sleeping sickness. PLoS Negl Trop Dis. 2012;6(10):e1859. doi: 10.1371/journal.pntd.0001859. Epub 2012 Oct 25. PMID 23145192
- [Background] Ngay Lukusa I, Van Reet N, Mumba Ngoyi D, Miaka EM, Masumu J, Patient Pyana P, Mutombo W, Ngolo D, Kobo V, Akwaso F, Ilunga M, Kaninda L, Mutanda S, Muamba DM, Valverde Mordt O, Tarral A, Rembry S, Buscher P, Lejon V. Trypanosome SL-RNA detection in blood and cerebrospinal fluid to demonstrate active gambiense human African trypanosomiasis infection. PLoS Negl Trop Dis. 2021 Sep 17;15(9):e0009739. doi: 10.1371/journal.pntd.0009739. eCollection 2021 Sep. PMID 34534223
- [Background] Van Reet N, Patient Pyana P, Dehou S, Bebronne N, Deborggraeve S, Buscher P. Single nucleotide polymorphisms and copy-number variations in the Trypanosoma brucei repeat (TBR) sequence can be used to enhance amplification and genotyping of Trypanozoon strains. PLoS One. 2021 Oct 25;16(10):e0258711. doi: 10.1371/journal.pone.0258711. eCollection 2021. PMID 34695154
- [Background] Simarro PP, Sima FO, Mir M, Mateo MJ, Roche J. [Control of human African trypanosomiasis in Luba in equatorial Guinea:evaluation of three methods]. Bull World Health Organ. 1991;69(4):451-7. PMID 1934239
- [Background] Buscher P, Mertens P, Leclipteux T, Gilleman Q, Jacquet D, Mumba-Ngoyi D, Pyana PP, Boelaert M, Lejon V. Sensitivity and specificity of HAT Sero-K-SeT, a rapid diagnostic test for serodiagnosis of sleeping sickness caused by Trypanosoma brucei gambiense: a case-control study. Lancet Glob Health. 2014 Jun;2(6):e359-63. doi: 10.1016/S2214-109X(14)70203-7. Epub 2014 May 9. PMID 25103304
- [Background] Camara O, Camara M, Falzon LC, Ilboudo H, Kabore J, Compaore CFA, Fevre EM, Buscher P, Bucheton B, Lejon V. Performance of clinical signs and symptoms, rapid and reference laboratory diagnostic tests for diagnosis of human African trypanosomiasis by passive screening in Guinea: a prospective diagnostic accuracy study. Infect Dis Poverty. 2023 Mar 20;12(1):22. doi: 10.1186/s40249-023-01076-1. PMID 36941656
- [Background] Compaore CFA, Kabore J, Ilboudo H, Thomas LF, Falzon LC, Bamba M, Sakande H, Kone M, Kaba D, Bougouma C, Adama I, Amathe O, Belem AMG, Fevre EM, Buscher P, Lejon V, Jamonneau V. Monitoring the elimination of gambiense human African trypanosomiasis in the historical focus of Batie, South-West Burkina Faso. Parasite. 2022;29:25. doi: 10.1051/parasite/2022024. Epub 2022 May 11. PMID 35543528
- [Derived] Nicco E, Lejon V, Mwamba Miaka E, Mumba D, Mpanya A, Kambo C, Ngolo D, Mutombo W, Hugonnet S, Rembry S, Tipple C, Inocencio Da Luz R, Snijders R, Vander Kelen C, Roge S, Van Reet N, Tarral A, Verle P, Hasker E. The STROGHAT study protocol: An intervention study to evaluate safety, effectiveness and feasibility of treating gambiense HAT seropositive subjects with acoziborole. Open Res Eur. 2025 Jan 24;5:23. doi: 10.12688/openreseurope.19077.1. eCollection 2025. PMID 40191624